## CONSENT FORM FOR TEACHER PARTICIPATION IN HUMAN RESEARCH AT MONTANA STATE UNIVERSITY

**PROJECT TITLE**: A Trauma-Informed Intervention for Positive Youth Development and Teacher Wellness in Rural Montana

INVESTIGATOR: Lauren Davis, Assistant Professor, Montana State University

RATIONALE FOR THE RESEARCH: We would like to invite you to participate in a research project to learn about how certain activities might help relieve your stress and improve your quality of life and job satisfaction. We are asking for your help because we don't know very much about how to best support teacher wellbeing, which in turn supports student wellbeing and achievement. Participation in this study is completely voluntary. If you agree to participate in our study, we are going to ask you to answer some questions about your stress levels, career satisfaction, and overall wellbeing before and after this 6-week program. We want to know if certain activities help reduce your stress—specifically, yoga. Here's what the program will look like:

\*Yoga: Each session will highlight deep breathing, mindful movement, and stress relief. Sessions will begin with goal-setting, will move into the physical practice, and will end with a peaceful reflection that will help you feel less stressed. This program will take place twice weekly, online and synchronously, for 6 weeks. You may have students participating in a student-version of this program at the same time as you during their physical education class and/or online.

At the end of the program, we may ask you if you feel like you are less burned out at work, if you feel less stressed out, or if you feel happier or less anxious. In order to measure your stress levels, your stress hormone (cortisol) levels will be tested throughout the program through a collected saliva (spit) sample; you can learn more about the procedure for this safe, non-invasive process here:

https://www.nationwidechildrens.org/family-resources-education/health-wellness-and-safety-resources/helping-hands/saliva-cortisol-test-collection-guidelines. We will also be measuring your resting heart rate variability with a sensor at three points during the study. As an incentive for your participation, if you complete all of the study activities, you will be eligible to receive payment for each class session in the form of a gift card, as well as a gift card for completing all surveys. Because of our budget, we are limiting participation to the first 40 teachers to sign up for the study. You can ask questions about the details of study at any time. If you decide at any time not to continue participating, then you won't be a part of the study.

The questions we will ask are only about what you think and feel before and after the study, which will take place for 6 weeks. There are no right or wrong answers; this is not a test. We will also ask you to write down and share with your reactions to the yoga sessions in an online journal each week so we can learn what was helpful to you in this study

**PROCEDURES:** Participation is voluntary. If you agree to participate, the confidential survey data you provide will be used in the study, and your responses will be kept anonymous. You will also be eligible for participation incentives (see below).

RISKS OF PARTICIPATION: It is possible that the program may bring up strong feelings for you; it's important for you to know your own limits and take care of yourself during the program. If you ask or if you need it, we will give you information for where you can find extra support. Some examples are:

- Talking with someone who you can trust
- Calling 911, your doctor or other healthcare provider

- Going to an Emergency Room Calling 1-800-273-TALK (8255) to talk with a crisis worker for free
- Texting 741741 to text with a counselor for free
- Visiting NowMattersNow.org to learn skills for dealing with thoughts of suicide

BENEFITS OF PARTICIPATION: Importantly, there are also potential benefits to being part of the study. You may have reductions in severity of depression and/or anxiety as well as improvements in overall behavioral health and well-being. Additional benefits for participants may be improved sleep, improved social skills, improved emotion regulation, and improvements in career satisfaction and/or burnout.

CONFIDENTIALITY: All research information will be kept confidential. All information will be kept in a secure platform that is accessible only to the researchers by password and institutional credentials. This information will be saved as long as it is scientifically useful; typically, such information is kept for five years after publication of the results. Results from this study may be presented at professional meetings and in publications. You will not be identified individually.

COMPENSATION: Teacher incentives for narticination in the study will be in the

| form of a gift card at the rate of \$15 per yoga clanditional gift cards of \$50 will be offered for conduring the study. | ass (limit of 12 classes total). |
|---|---|
| I, | |
| understand this consent form. I sign it freely and<br>permission for my participation in this study and<br>the study at a later time. I have received a copy | I understand that I may withdraw from of this consent form. |
| | Signature of Participant |
| Date | |

Contact Information: Dr. Lauren Davis (Principal Investigator) Montana State University Lauren.davis6@montana.edu 406-994-7424

Note: This form is a requirement of Montana State University's Institutional Review Board (IRB). An IRB is an administrative body established to protect the rights and welfare of human research subjects recruited to participate in research activities conducted by faculty members of Montana State University. The IRB is charged with the responsibility of reviewing, prior to its initiation, all research involving human participants. The IRB is concerned with protecting the welfare, rights, and privacy of human subjects and has the authority to approve, disapprove, monitor, and require modifications in all research activities that fall within its jurisdiction as specified by both the federal regulations and institutional policy. If you have any questions regarding this proposed project, their contact information is listed below; please don't hesitate to reach out to them with any concerns. Montana State University Institutional Review Board Mark Quinn, Chair P.O. Box 173610 Bozeman, MT 59717